CLINICAL TRIAL: NCT02704091
Title: Efficacy of Diosmectite (Smecta®) in the Symptomatic Treatment of Acute Diarrhoea in Adults. A Multicentre, Randomized, Double Blind Placebo Controlled, Parallel, Groups Study
Brief Title: Efficacy of Diosmectite (Smecta®) in the Symptomatic Treatment of Acute Diarrhoea in Adults
Acronym: ADIASE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F-FR-00250-105; 2015-001138-10 (EudraCT Number)
Record Dates: First submitted 2016-03-04; First posted 2016-03-09 (Estimated); Results first posted 2020-04-24 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Acute Diarrhoea
MeSH Terms: interventions — smecta

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smecta (Active Comparator): 2 sachets, three times a day (TID), during 5 to 9 days
  Interventions: Drug: Smecta
- Smecta placebo (Placebo Comparator): 2 sachets of placebo, TID, during 5 to 9 days
  Interventions: Drug: Smecta placebo

INTERVENTIONS:
Drug: Smecta
  Other Names: Diosmectite Beaufour
  Arms: Smecta
Drug: Smecta placebo
  Arms: Smecta placebo

SUMMARY:
The purpose of the study is to demonstrate that diosmectite efficacy is superior to placebo regarding time to recovery of an acute diarrhoea episode presumed of infectious origin in adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent prior to any study related procedures
* Male or female subject (outpatient) legally considered as an adult (age of majority). In Czech Republic, the upper limit of age will be 70 years inclusive. In Egypt, the upper limit of age will be 60 years inclusive.
* Subject has a diagnosis of acute diarrhoea presumed of infectious origin, defined as the passage of 3 or more unformed loose or watery stools (rated according to the Bristol scale) per day within the last 48 hours without associated alarm symptoms
* Subject has, usually, normal bowel habits (Rome III criteria), i.e. at least 3 stools per week and no more than 3 stools per day
* Subject must be willing and able to comply with study restrictions and willing to return to the clinic for the follow up evaluation(s) as specified in the protocol.

Exclusion criteria related to the acute diarrhoea episode:

* At least one of the following alarm symptoms

  * Bloody diarrhoea*,
  * pus in the stools*,
  * fever ≥38°C*,
  * moderate or severe dehydration according to World Health Organisation (WHO) definition, requiring intravenous (IV) rehydration*,
  * repeated vomiting*,
  * persistent abdominal pain* *These symptoms are considered as alarm symptoms
* other episode of acute watery diarrhoea within the previous 30 days,
* persistent diarrhoea, defined as acutely starting episode of diarrhoea lasting more than 14 days,
* history of chronic diarrhoea (Rome III criteria); i.e. 3 or more loose or watery stools per day for at least 12 weeks, consecutive or not, in the preceding 12 months,
* traveller's diarrhoea defined as a diarrhoeal episode due to contamination experienced by subjects having travelled in at risk countries, or coming from abroad and experiencing locally an acute diarrhoea episode, occurring usually within the first 2 weeks of the stay in a foreign environment.

Exclusion criteria related to drugs:

* Diarrhoea suspected to be induced by drug for example:

  * antibiotic therapy, including Clostridium difficile-induced diarrhoea, within 1 week before entry in the study,
  * laxative agent
  * thyroid hormone (at a nonstabilised dosing),
  * intake of other prohibited drugs (as specified in the protocol)
* anti-diarrhoeal agent intake during the last month,
* any subject requiring repeated intake of a drug with a narrow therapeutic margin (as specified in the protocol),
* history of hypersensitivity to diosmectite or its excipients or placebo components,
* subject likely to require treatment during the study with drugs that are not permitted by the study protocol (for example, antibiotic agent, anti-diarrhoeal agent, antiemetic drug, antispasmodic drug),
* use of any investigational medication within the last 30 days before entering this study,
* subject who previously entered in a clinical study within the past 30 days.

Other digestive exclusion criteria:

* History of gastric or intestinal resection, vagotomy,
* known digestive malabsorption disease, including coeliac disease
* known lactose intolerance,
* any suspicion of abdominal surgery need,
* known inflammatory bowel disease.

Other exclusion criteria:

* Known Human immunodeficiency virus (HIV) positive status,
* known or suspected immunosuppression,
* known severe renal insufficiency (including e-GFR not less than 45 mL/min) or hepatic insufficiency,
* known endocrine disease or Type II Diabetes Mellitus with HBA1c more than 8,5% or insulin-dependent diabetes,
* history of, or known current, problems with alcohol abuse and/or known drug addiction (cocaine, heroin, hashish…),
* previous enrolment in this study,
* any mental condition rendering the subject unable to understand the nature, scope and possible consequences of the study, and/or evidence of an uncooperative attitude.
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 858 (Actual)
Dates: Start 2016-03-17 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (70):
- Algeria (14):
  - Cabinet privé, Coopératives El MOSTAKBAL, BIRKHADEM, Algiers
  - CHU Beni Messous, Algiers
  - CHU Mustapha, Algiers
  - Polyclinique d'el Achour, Algiers
  - Polyclinique de Baba Hassen, Algiers
  - Cabinet privé, 29 avenue amara Youcef, Blida
  - EPH Blida, Blida
  - EPH EL Afroun, Blida
  - EPH Bologhine, Bologhine
  - Cabinet privé, cité des 408 lgmts Bt3, Boumerdas
  - CHU BEN BADIS Constantine, Constantine
  - Polyclinique de Dély Brahim, Deli Ibrahim
  - Polyclinique DRARIA, Draria
  - CHU Oran, Oran
- Czechia (14):
  - Ordinace PL pro dospělé, Prague, Karlín
  - Ordinace PL pro dospělé, Prague, Nusle
  - Ordinace PL pro dospělé, Prague, Vysočany
  - Ordinace PL pro dospělé, Čáslav
  - OPL, spol. s r.o., Hrochův Týnec
  - Ordinace PL pro dospělé, Kladno
  - Ordinace PL pro dospělé, Poliklinika přízemí, Nerudova, Kralupy nad Vltavou
  - AK Medipraktik, s.r.o, Orlová
  - MUDr. Alena Břeňová - PL pro dospělé, Pardubice
  - Ordinace Bělehradská s.r.o, Prague
  - Ordinace PL pro dospělé, Prague
  - Ordinace PL pro dospělé, Praha 6, 2.patro
  - Praktický lékař Radotín, s.r.o., Radotín
  - Ordinace PL pro dospělé, Vrchlabí
- Egypt (7):
  - Clinical Research Center, Alexandria
  - Ain Shams University Hospitals, Cairo
  - Air Force Specialized Hospital, Cairo
  - Al Hussein University Hospital, Cairo
  - Badr University Hospital, Cairo
  - Cairo University, Cairo
  - Tanta University, Tanta
- Hammoud Hospital University Medical Center, Sidon, Lebanon
- Poland (15):
  - Komisji Edukacji Narodowej 3B lok. 1, Bialystok
  - Cermed, Bialystok
  - KLIMED, Bychawa
  - Indywidualna Specjalistyczna Praktyka Lekarska Roman Spyra, Katowice
  - MEKMED S.C. Przychodnia Lekarska NZOZ, Katowice
  - Lekarska Spółka Partnerska Familia T S A Gugała, Kozienice
  - Praktyka Lekarzy Rodzinnych NZOZ, Krakow
  - Niepubliczny Zakład Opieki Zdrowotnej Ugorek sp. z o.o., Krakow
  - Niepubliczny Zakład Opieki Zdrowotnej Centrum Zdrowia i Profilaktyki "Dąbie" spółka z o.o., Krakow
  - Niepubliczny Zakład Opieki Zdrowotnej Praktyka Lekarza Rodzinnego "Eskulap" spółka z o.o., Lublin
  - NZOZ Primed, Malbork
  - Solumed Research Site, Poznan
  - Centrum Medyczne Pratia S.A, Warsaw
  - PrzychodniaLekarska ORLIK Sp. z o.o, Warsaw
  - KLIMED, Łomża
- Tunisia (19):
  - CSB Zouhour, Ben Arous
  - Hôpital Régional de Ben Arous, Ben Arous
  - Centre intermédiaire de Santé de Base, La Marsa
  - Hôpital des Forces de Sécurité Intérieure, La Marsa
  - CSB Hedi Chaker, Sousse
  - Hôpital Universitaire Salhoul, Sousse
  - CSB Akouda, Sousse
  - CSB Sidi Bou Ali, Sousse
  - CSB Zouhour, Sousse
  - CSB Nager, Sousse
  - CSB Riadh, Sousse
  - CSB Oued Blibène, Sousse
  - CSB Kalaa Kébira, Sousse
  - CSB Zaouia, Sousse
  - Centre de santé de base Bab Laasal, Tunis
  - Hopital Militaire Principal d'instructions de Tunis, Tunis
  - Centre de santé de base Ras Tabia, Tunis
  - Centre de santé de base Ksar Said, Tunis
  - Centre de santé de base Ibn Khaldoun, Tunis

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled adult participants with a recent episode of acute diarrhoea presumed of infectious origin, defined as the passage of 3 or more unformed (loose or watery) stools per day without alarm symptoms within the first 48 hours. Participants were randomised at 62 study centres in Algeria, Czech Republic, Egypt, Lebanon, Poland and Tunisia.
Pre-assignment Details: 858 participants were randomised, of which 853 were included in the analysis and 5 were excluded due to invalid consent. Only participants included in the analysis are presented in the participant flow. Participants received a diary evaluation booklet (DEB) to record each stool plus consistency on a daily basis from inclusion until end of study.
Groups:
- Diosmectite: Participants received diosmectite as 2 sachets, three times a day (TID) (2 sachets in the morning, 2 sachets at mid-day, and 2 sachets in the evening). Each sachet was taken in half a glass of water.
  The mandatory treatment period was from Day 1 to Day 4 or Day 5 (with a minimum of 24 sachets taken within 4 or 5 days). Treatment could continue from Day 5 up to Day 8 or 9 (with a maximum of 48 sachets taken within 8 or 9 days).
- Placebo: Participants received matching placebo as 2 sachets, TID (2 sachets in the morning, 2 sachets at mid-day, and 2 sachets in the evening). Each sachet was taken in half a glass of water.
  The mandatory treatment period was from Day 1 to Day 4 or Day 5 (with a minimum of 24 sachets taken within 4 or 5 days). Treatment could continue from Day 5 up to Day 8 or 9 (with a maximum of 48 sachets taken within 8 or 9 days).
Period: Overall Study
Arm/Group | Diosmectite | Placebo
Started | 430 | 423
Completed | 402 | 400
Not Completed | 28 | 23
Not completed — Adverse Event | 4 | 3
Not completed — Protocol Violation | 5 | 3
Not completed — Consent withdrawn | 4 | 4
Not completed — Lost to Follow-up | 13 | 5
Not completed — Other | 2 | 8

BASELINE CHARACTERISTICS:
Population: The Intention-To-Treat (ITT) population included all randomised participants, analysed according to the arm to which they were randomised, except for those excluded from the analysis.
Groups:
- Diosmectite: Participants received diosmectite as 2 sachets, TID (2 sachets in the morning, 2 sachets at mid-day, and 2 sachets in the evening). Each sachet was taken in half a glass of water.
  The mandatory treatment period was from Day 1 to Day 4 or Day 5 (with a minimum of 24 sachets taken within 4 or 5 days). Treatment could continue from Day 5 up to Day 8 or 9 (with a maximum of 48 sachets taken within 8 or 9 days).
Arm/Group | Diosmectite | Placebo | Total Title
Number analyzed (Participants) | 430 | 423 | 853
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (14.5) | 38.6 (14.2) | 39.1 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 232 | 241 | 473
  Male | 198 | 182 | 380
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Time to Recovery
Description: Time to recovery was defined as the time from the first study treatment intake recorded in the electronic case report form (eCRF) to the first formed stool followed by a non-watery stool, recorded in the DEB. Results are presented as median time to recovery, calculated using the Kaplan-Meier technique. Participants prematurely withdrawn without recovery or ending the study without recovery were censored (not responders) at the date/time of their last stool as recorded in the DEB. Participants who had not filled in the DEB (i.e. no post-baseline evaluation of stools) were censored at the date/time of their first study treatment intake (or the randomisation date/time if not administered).
Time Frame: From randomisation (Day 1) up to Day 9
Population: The ITT population included all randomised participants (except for those excluded from the analysis), analysed according to the arm to which they were randomised.
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Diosmectite | Placebo
Number analyzed (Participants) | 430 | 423
Hours | 66.0 [53.7 to 71.0] | 68.6 [57.5 to 77.8]
Statistical Analysis 1: Comparison: Diosmectite vs Placebo; The primary analysis tested the equality of time to recovery between the 2 treatment groups, applying the 2-sided Gehan-Wilcoxon test (α=5%); Test type: Superiority — The following Null-hypothesis was tested: H0: λA(t) = λB (t) versus H1: λA(t) ≠ λB (t), where λ(t) represents the hazard at time t, A=diosmectite and B=placebo; p = 0.2524, Wilcoxon-Gehan test

2. Secondary Outcome: Time From Diarrhoea Onset to Recovery
Description: The event of diarrhoea onset (i.e. loose or watery stool) was recorded in the eCRF and the event of recovery (i.e. first formed stool followed by a non-watery stool) was recorded in the DEB. Results are presented as median time from diarrhoea onset to recovery, calculated using the Kaplan-Meier technique. Participants prematurely withdrawn without recovery or ending the study without recovery were censored (not responders) at the date/time of their last stool as recorded in the DEB. Participants who had not filled in the DEB (i.e. no post-baseline evaluation of stools) were censored at the date/time of their first study treatment intake (or the randomisation date/time if not administered).
Time Frame: From randomisation (Day 1) up to Day 9
Population: The ITT population included all randomised participants (with the exception of those excluded from the analysis), analysed according to the arm to which they were randomised. Only participants with data available were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Diosmectite | Placebo
Number analyzed (Participants) | 429 | 423
Hours | 91.0 [82.5 to 107.0] | 92.2 [84.2 to 102.8]
Statistical Analysis 1: Comparison: Diosmectite vs Placebo; Comparison between the 2 treatment groups for time from diarrhoea onset to recovery, analysed using the Gehan-Wilcoxon test; Test type: Superiority; p = 0.3511, Gehan-Wilcoxon test

3. Secondary Outcome: Time From Diarrhoea Onset to First Formed Stool
Description: The event of diarrhoea onset (i.e. loose or watery stool) was recorded in the eCRF and the event of first formed stool was recorded in the DEB. Results are presented as median time from diarrhoea onset to first formed stool, calculated using the Kaplan-Meier technique. Participants prematurely withdrawn with no formed stool or ending the study with no formed stool were censored at the date/time of their last stool as recorded in the DEB. Participants who had not filled in the DEB (i.e. no post-baseline evaluation of stools) were censored at the date/time of their first study treatment intake (or the randomisation date/time if not administered).
Time Frame: From randomisation (Day 1) up to Day 9
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Diosmectite | Placebo
Number analyzed (Participants) | 429 | 423
Hours | 84.3 [77.5 to 94.2] | 84.6 [79.8 to 91.0]
Statistical Analysis 1: Comparison: Diosmectite vs Placebo; Comparison between the 2 treatment groups for time from diarrhoea onset to first formed stool, analysed using the Gehan-Wilcoxon test; Test type: Superiority; p = 0.7285, Gehan-Wilcoxon test

4. Secondary Outcome: Time From the First Study Treatment Intake to the Last Watery Stool
Description: The event of first study treatment intake was recorded in the eCRF and the event of last watery stool was recorded in the DEB. Results are presented as median time from first study treatment intake to last watery stool, calculated using the Kaplan-Meier technique. Participants prematurely withdrawn with no watery stool or ending the study with no watery stool were censored at the date/time of their last stool as recorded in the DEB. Participants who had not filled in the DEB (i.e. no post-baseline evaluation of stools) were censored at the date/time of their first study treatment intake (or the randomisation date/time if not administered).
Time Frame: From randomisation (Day 1) up to Day 9
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Diosmectite | Placebo
Number analyzed (Participants) | 430 | 423
Hours | 56.2 [44.6 to 66.2] | 60.0 [52.8 to 68.8]
Statistical Analysis 1: Comparison: Diosmectite vs Placebo; Comparison between the 2 treatment groups for time from first study treatment intake to last watery stool, analysed using the Gehan-Wilcoxon test; Test type: Superiority; p = 0.1807, Gehan-Wilcoxon test

5. Secondary Outcome: Number of Stools, Per 12-Hour Period
Description: Number of stools, per 12-hour period, was recorded in the DEB.
Time Frame: From randomisation (Day 1) up to Day 9
Population: The ITT population included all randomised participants (with the exception of those excluded from the analysis), analysed according to the arm to which they were randomised. Only participants with data available at each specified time point were included in the analysis.
Measure: Median (Full Range); unit: Stools
Arm/Group | Diosmectite | Placebo
Number analyzed (Participants) | 413 | 412
Stools
  0 - 12 hours | 3.0 [0 to 11] | 3.0 [0 to 14]
  12 - 24 hours: number analyzed (Participants) | 407 | 411
  12 - 24 hours | 2.0 [0 to 7] | 2.0 [0 to 7]
  24 - 36 hours: number analyzed (Participants) | 402 | 407
  24 - 36 hours | 1.0 [0 to 8] | 2.0 [0 to 19]
  36 - 48 hours: number analyzed (Participants) | 396 | 400
  36 - 48 hours | 1.0 [0 to 7] | 1.0 [0 to 6]
  48 - 60 hours: number analyzed (Participants) | 386 | 391
  48 - 60 hours | 1.0 [0 to 7] | 1.0 [0 to 9]
  60 - 72 hours: number analyzed (Participants) | 373 | 383
  60 - 72 hours | 1.0 [0 to 6] | 1.0 [0 to 7]
  72 - 84 hours: number analyzed (Participants) | 320 | 329
  72 - 84 hours | 1.0 [0 to 12] | 1.0 [0 to 7]
  84 - 96 hours: number analyzed (Participants) | 269 | 264
  84 - 96 hours | 1.0 [0 to 6] | 1.0 [0 to 7]
  96 - 108 hours: number analyzed (Participants) | 191 | 174
  96 - 108 hours | 1.0 [0 to 5] | 1.0 [0 to 7]
  108 - 120 hours: number analyzed (Participants) | 151 | 143
  108 - 120 hours | 1.0 [0 to 5] | 1.0 [0 to 6]
  120 - 132 hours: number analyzed (Participants) | 109 | 120
  120 - 132 hours | 1.0 [0 to 4] | 1.0 [0 to 6]
  132 - 144 hours: number analyzed (Participants) | 95 | 109
  132 - 144 hours | 1.0 [0 to 6] | 1.0 [0 to 4]
  144 - 156 hours: number analyzed (Participants) | 75 | 100
  144 - 156 hours | 1.0 [0 to 4] | 1.0 [0 to 6]
  156 - 168 hours: number analyzed (Participants) | 57 | 80
  156 - 168 hours | 1.0 [0 to 4] | 1.0 [0 to 5]
  168 - 180 hours: number analyzed (Participants) | 42 | 60
  168 - 180 hours | 1.0 [0 to 5] | 1.0 [0 to 4]
  180 - 192 hours: number analyzed (Participants) | 32 | 44
  180 - 192 hours | 1.0 [0 to 5] | 1.0 [0 to 5]
  192 - 204 hours: number analyzed (Participants) | 17 | 16
  192 - 204 hours | 1.0 [1 to 4] | 1.0 [0 to 4]
  204 - 216 hours: number analyzed (Participants) | 0 | 1
  204 - 216 hours |  | 1.0 [1 to 1]
Statistical Analysis 1: Comparison: Diosmectite vs Placebo; Comparison between the 2 treatment groups for number of stools for the overall time period, based on an analysis of covariance (ANCOVA) method for repeated measurements. The model included the number of stools 24 hours before randomisation (baseline) as covariate, treatment, time point (12-hour period), the treatment by time point interaction as fixed effects and participant as random effect; Test type: Superiority; p = 0.4294, ANCOVA; Least Squares (LS) Mean Difference = -0.04, 95% CI 2-sided [-0.15 to 0.07]

6. Secondary Outcome: Number of Watery Stools, Per 12-Hour Period
Description: Number of watery stools, per 12-hour period, was recorded in the DEB.
Time Frame: From randomisation (Day 1) up to Day 9
Population: as for outcome 5
Measure: Median (Full Range); unit: Stools
Arm/Group | Diosmectite | Placebo
Number analyzed (Participants) | 413 | 412
Stools
  0 - 12 hours | 3.0 [0 to 11] | 3.0 [0 to 14]
  12 - 24 hours: number analyzed (Participants) | 407 | 411
  12 - 24 hours | 1.0 [0 to 7] | 1.0 [0 to 7]
  24 - 36 hours: number analyzed (Participants) | 402 | 407
  24 - 36 hours | 0.0 [0 to 8] | 1.0 [0 to 19]
  36 - 48 hours: number analyzed (Participants) | 396 | 400
  36 - 48 hours | 0.0 [0 to 7] | 0.0 [0 to 6]
  48 - 60 hours: number analyzed (Participants) | 386 | 391
  48 - 60 hours | 0.0 [0 to 7] | 0.0 [0 to 9]
  60 - 72 hours: number analyzed (Participants) | 373 | 383
  60 - 72 hours | 0.0 [0 to 6] | 0.0 [0 to 7]
  72 - 84 hours: number analyzed (Participants) | 320 | 329
  72 - 84 hours | 0.0 [0 to 10] | 0.0 [0 to 7]
  84 - 96 hours: number analyzed (Participants) | 269 | 264
  84 - 96 hours | 0.0 [0 to 6] | 0.0 [0 to 7]
  96 - 108 hours: number analyzed (Participants) | 191 | 174
  96 - 108 hours | 0.0 [0 to 5] | 0.0 [0 to 7]
  108 - 120 hours: number analyzed (Participants) | 151 | 143
  108 - 120 hours | 0.0 [0 to 5] | 0.0 [0 to 6]
  120 - 132 hours: number analyzed (Participants) | 109 | 120
  120 - 132 hours | 0.0 [0 to 4] | 0.0 [0 to 5]
  132 - 144 hours: number analyzed (Participants) | 95 | 109
  132 - 144 hours | 0.0 [0 to 6] | 0.0 [0 to 4]
  144 - 156 hours: number analyzed (Participants) | 75 | 100
  144 - 156 hours | 0.0 [0 to 3] | 0.0 [0 to 5]
  156 - 168 hours: number analyzed (Participants) | 57 | 80
  156 - 168 hours | 0.0 [0 to 4] | 0.0 [0 to 5]
  168 - 180 hours: number analyzed (Participants) | 42 | 60
  168 - 180 hours | 0.0 [0 to 5] | 0.0 [0 to 4]
  180 - 192 hours: number analyzed (Participants) | 32 | 44
  180 - 192 hours | 0.0 [0 to 5] | 0.0 [0 to 5]
  192 - 204 hours: number analyzed (Participants) | 17 | 16
  192 - 204 hours | 0.0 [0 to 4] | 0.0 [0 to 3]
  204 - 216 hours: number analyzed (Participants) | 0 | 1
  204 - 216 hours |  | 0.0 [0 to 0]
Statistical Analysis 1: Comparison: Diosmectite vs Placebo; Comparison between the 2 treatment groups for number of watery stools for the overall time period, based on an ANCOVA method for repeated measurements. The model included the number of watery stools 24 hours before randomisation (baseline) as covariate, treatment, time point (12-hour period), the treatment by time point interaction as fixed effects and participant as random effect; Test type: Superiority; p = 0.0465, ANCOVA; LS Mean Difference = -0.12, 95% CI 2-sided [-0.24 to -0.00]

7. Secondary Outcome: Percentage of Participants With Associated Symptoms, Per 12-Hour Period
Description: Percentage of participants with associated symptoms (at least 1 symptom of nausea, vomiting, abdominal pain or anal irritation) per 12-hour period is presented. Nausea, vomiting, abdominal pain and anal irritation were recorded in the DEB.
Time Frame: From randomisation (Day 1) up to Day 9
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Diosmectite | Placebo
Number analyzed (Participants) | 430 | 423
Percentage of participants
  0 - 12 hours: number analyzed (Participants) | 400 | 390
  0 - 12 hours | 76.3 | 76.4
  12 - 24 hours: number analyzed (Participants) | 395 | 395
  12 - 24 hours | 67.1 | 64.6
  24 - 36 hours | 56.2 | 54.2
  36 - 48 hours: number analyzed (Participants) | 395 | 395
  36 - 48 hours | 44.8 | 45.6
  48 - 60 hours: number analyzed (Participants) | 392 | 395
  48 - 60 hours | 34.9 | 35.4
  60 - 72 hours: number analyzed (Participants) | 376 | 379
  60 - 72 hours | 28.7 | 28.8
  72 - 84 hours: number analyzed (Participants) | 370 | 381
  72 - 84 hours | 24.3 | 22.0
  84 - 96 hours: number analyzed (Participants) | 329 | 345
  84 - 96 hours | 21.6 | 20.6
  96 - 108 hours: number analyzed (Participants) | 228 | 242
  96 - 108 hours | 20.6 | 24.0
  108 - 120 hours: number analyzed (Participants) | 177 | 173
  108 - 120 hours | 18.6 | 24.9
  120 - 132 hours: number analyzed (Participants) | 136 | 136
  120 - 132 hours | 18.4 | 27.9
  132 - 144 hours: number analyzed (Participants) | 103 | 117
  132 - 144 hours | 12.6 | 21.4
  144 - 156 hours: number analyzed (Participants) | 86 | 104
  144 - 156 hours | 10.5 | 19.2
  156 - 168 hours: number analyzed (Participants) | 71 | 87
  156 - 168 hours | 8.5 | 16.1
  168 - 180 hours: number analyzed (Participants) | 58 | 76
  168 - 180 hours | 8.6 | 11.8
  180 - 192 hours: number analyzed (Participants) | 49 | 61
  180 - 192 hours | 8.2 | 9.8
  192 - 204 hours: number analyzed (Participants) | 31 | 38
  192 - 204 hours | 9.7 | 10.5
  204 - 216 hours: number analyzed (Participants) | 17 | 20
  204 - 216 hours | 5.9 | 0.0

8. Secondary Outcome: Abdominal Pain Intensity Scores, Per 12-Hour Period
Description: Abdominal pain intensity per 12-hour period was recorded in the DEB. Abdominal pain intensity was rated with a 5-point ordinal scale: 0 = absent, 1= mild, 2 =moderate, 3 = severe, 4= very severe. Higher scores indicate a worse outcome. The median abdominal pain intensity score for each 12-hour period is presented.
Time Frame: From randomisation (Day 1) up to Day 9
Population: as for outcome 5
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Diosmectite | Placebo
Number analyzed (Participants) | 430 | 423
Scores on a scale
  0 - 12 hours: number analyzed (Participants) | 384 | 377
  0 - 12 hours | 1.0 [0 to 4] | 1.0 [0 to 4]
  12 - 24 hours: number analyzed (Participants) | 382 | 379
  12 - 24 hours | 1.0 [0 to 4] | 1.0 [0 to 4]
  24 - 36 hours | 0.0 [0 to 4] | 0.0 [0 to 4]
  36 - 48 hours: number analyzed (Participants) | 382 | 380
  36 - 48 hours | 0.0 [0 to 4] | 0.0 [0 to 4]
  48 - 60 hours: number analyzed (Participants) | 381 | 380
  48 - 60 hours | 0.0 [0 to 4] | 0.0 [0 to 4]
  60 - 72 hours: number analyzed (Participants) | 368 | 366
  60 - 72 hours | 0.0 [0 to 4] | 0.0 [0 to 4]
  72 - 84 hours: number analyzed (Participants) | 362 | 369
  72 - 84 hours | 0.0 [0 to 4] | 0.0 [0 to 4]
  84 - 96 hours: number analyzed (Participants) | 319 | 336
  84 - 96 hours | 0.0 [0 to 4] | 0.0 [0 to 4]
  96 - 108 hours: number analyzed (Participants) | 220 | 233
  96 - 108 hours | 0.0 [0 to 3] | 0.0 [0 to 4]
  108 - 120 hours: number analyzed (Participants) | 171 | 171
  108 - 120 hours | 0.0 [0 to 3] | 0.0 [0 to 4]
  120 - 132 hours: number analyzed (Participants) | 133 | 133
  120 - 132 hours | 0.0 [0 to 4] | 0.0 [0 to 4]
  132 - 144 hours: number analyzed (Participants) | 101 | 113
  132 - 144 hours | 0.0 [0 to 2] | 0.0 [0 to 4]
  144 - 156 hours: number analyzed (Participants) | 86 | 104
  144 - 156 hours | 0.0 [0 to 3] | 0.0 [0 to 4]
  156 - 168 hours: number analyzed (Participants) | 67 | 86
  156 - 168 hours | 0.0 [0 to 3] | 0.0 [0 to 4]
  168 - 180 hours: number analyzed (Participants) | 55 | 75
  168 - 180 hours | 0.0 [0 to 3] | 0.0 [0 to 4]
  180 - 192 hours: number analyzed (Participants) | 45 | 60
  180 - 192 hours | 0.0 [0 to 2] | 0.0 [0 to 4]
  192 - 204 hours: number analyzed (Participants) | 29 | 38
  192 - 204 hours | 0.0 [0 to 4] | 0.0 [0 to 4]
  204 - 216 hours: number analyzed (Participants) | 17 | 20
  204 - 216 hours | 0.0 [0 to 1] | 0.0 [0 to 0]

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events were collected from Day 1 until 7 days after the end of the study treatment, up to 16 days.
Description: The safety population included all randomised participants who received at least 1 dose of study treatment (except for those excluded from the analysis). Participants were analysed according to the actual treatment received.
Arm/Group | Diosmectite | Placebo
All-Cause Mortality (participants affected / at risk) | 0/430 | 0/421
Serious Adverse Events (participants affected / at risk) | 1/430 | 1/421
Other Adverse Events (participants affected / at risk) | 29/430 | 32/421
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diosmectite (N=430) | Placebo (N=421)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diosmectite (N=430) | Placebo (N=421)
Abdominal pain (Gastrointestinal disorders) | 9 (9) | 9 (9)
Anorectal discomfort (Gastrointestinal disorders) | 5 (5) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (4)
Proctalgia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anal pruritus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Arthritis salmonella (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Urethritis (Infections and infestations) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acrophobia (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor requires that reasonable opportunity be given to review the content and conclusions of any abstract, presentation, or paper before the material is submitted for publication or communicated. The sponsor will comment on the draft documents within the time period agreed in the contractual arrangements. Requested amendments will be incorporated by the author, provided they do not alter the scientific value of the material.

DOCUMENTS (2):
  • Study Protocol (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT02704091/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-15): https://cdn.clinicaltrials.gov/large-docs/91/NCT02704091/SAP_001.pdf